CLINICAL TRIAL: NCT01157858
Title: Everolimus Added to Long Acting Octreotide as a Volume Reducing Treatment of Polycystic Livers
Brief Title: Everolimus and LongActing Octreotide Trial in Polycystic Livers
Acronym: ELATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Joost Drenth, MD, PhD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995 ANLIIT
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Polycystic Liver Disease
Keywords: liver cyst
MeSH Terms: conditions — Polycystic liver disease | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus + octreotide LAR (Active Comparator): Octreotide LAR combined with everolimus
  Interventions: Drug: Everolimus; Drug: Octreotide LAR
- Octreotide LAR (Active Comparator): Octreotide LAR monotherapy
  Interventions: Drug: Octreotide LAR

INTERVENTIONS:
Drug: Everolimus — 2.5 mg every day orally
  Other Names: Afinitor
  Arms: Everolimus + octreotide LAR
Drug: Octreotide LAR — 40 mg every 28 days IM
  Other Names: Sandostatine LAR

SUMMARY:
The aim of this study is to reduce polycystic liver volume by treating with octreotide, whether or not combined with everolimus; to assess whether combination therapy of everolimus and octreotide gives a bigger reduction of polycystic liver volume than octreotide monotherapy.

DETAILED DESCRIPTION:
This is a single center randomized, open-label, parallel study comparing the safety and efficacy of everolimus-octreotide LAR treatment to monotherapy octreotide LAR in adult symptomatic patients with polycystic livers because of polycystic liver disease (PCLD).

We aim to include 44 patients affected by a polycystic liver either due to PCLD, 22 patients in the combination group and 22 patients in the mono therapy group.The duration of the trial will be 52 weeks. The treatment will be 48 weeks and the last control visit will take place four weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 < age ≤ 70 years
* Polycystic liver disease (PCLD), defined as ≥ 20 liver cysts
* Total liver volume must be at least 2500 mL
* Symptomatic defined as ECOG-PS ≥ 1 (see fig 3.1)38, and having at least three out of ten PCLD symptoms:
* Abdominal pain
* Abdominal distension
* Abdominal fullness
* Dyspnea
* Early satiety
* Back pain
* Nausea/vomiting
* Anorexia
* Weight loss
* Jaundice
* Informed consent, patients are willing and able to comply with the study drug regimen and all other study requirements

Exclusion Criteria:

* ADPKD patients
* Use of oral anticonceptives or estrogen supplementation
* Females who are pregnant or breast-feeding or patients of reproductive potential not employing an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to the administration of study medication.
* Intervention (aspiration or surgical intervention) within three months before baseline
* Treatment with somatostatin analogues within three months before baseline
* Patients with a kidney transplant
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of severe cardiac disease (eg, NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases). In addition, patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Symptomatic gallstones (octreotide decreases gall bladder volume)
* Hypercholesterolemia (fasting cholesterol > 8 mmol/l) or hypertriglyceridaemia (> 5 mmol/l) not controlled by lipid lowering therapy
* Granulocytopenia (white blood cell < 3,000/mm3) or thrombocytopenia (platelets < 100,000/mm3)
* Infection with hepatitis B, hepatitis C, HIV, TBC (in medical history)
* Mental illness that interferes with the patient ability to comply with the protocol
* Drug or alcohol abuse within one year of baseline
* Co-medication with strong inhibitor of CYP3A4 and or P-gp like voriconazole, ketoconazole, diltiazem, verapamil, erythromycin or with a strong CYP3A4 and or P-gp inductor like rifampicin
* Known hypersensitivity to everolimus or one of its excipients
* Enrolment in another clinical trial of an investigational agent while participating in this study
* Moderate or severe reaction on contrast in medical history
* Treatment with I131 during the course of the trial
* Use of metformin
* Morbus Kahler or Morbus Waldenstrom with excretion of light chains in urine in medical history
* Kidney dysfunction (MDRD-GFR < 60 ml/min/1.73m2 and ECC < 60 ml/min, calculated by the Cockcroft-Gault formula); in case of decreased body muscle mass, exact ECC is measured using serum and urine creatinine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Liver volume | at baseline and at 12 months
  change of total liver volume in terms of percentage from baseline to 12 months as determined by CT

SECONDARY OUTCOMES:
Symptoms | baseline and 12 months
  Change in symptoms, measured by GI-questionnaire
Quality of Life | baseline and 12 months
  Change in quality of life, measured by EuroQoL-questionnaire
Responders | baseline and 12 months
  Proportion of patients having any reduction in total liver volume after 12 months
Adverse events | During 12 months of treatment
  Adverse events that occur in these 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joost PH Drenth, MD, PhD, Principal Investigator — Radboud University Medical Center; Melissa Chrispijn, MD, Study Director — Radboud University Medical Center
Locations (1):
- Department of Gastroenterology and Hepatology, Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Chrispijn M, Drenth JP. Everolimus and long acting octreotide as a volume reducing treatment of polycystic livers (ELATE): study protocol for a randomized controlled trial. Trials. 2011 Nov 21;12:246. doi: 10.1186/1745-6215-12-246. PMID 22104015